CLINICAL TRIAL: NCT07347821
Title: Molecular Mechanisms Underlying Hip and Knee Osteoarthritis in Patients Undergoing Primary Elective Arthroplasty
Status: Recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: KB/129/2025
Record Dates: First submitted 2025-11-14; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-10

CONDITIONS: Total Hip Arthroplasty (THA); Total Knee Arthroplasty (TKA); Hip Osteoarthritis; Knee Osteoarthristis
Keywords: Total Knee Replacement; Total Hip Replacement; Trace Elements; Osteoarthritis; Cytokines; Oxidative Stress
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- patients undergoing primary total knee arthroplasty
- patients undergoing primary total hip arthroplasty

SUMMARY:
The aim of this observational study is to determine content of rare metals and other elements, along with the levels of selected immunological parameters, in the tissue of the hip or knee joint in the course of degenerative diseases. Determining potential disturbances in the levels or functions of these parameters may in the future contribute to improving treatment - for example, through supplementation of deficient metals or modulation at the immunological level. The main question it aims to answer is:

Are selected rare metals, trace elements and other selected immunological parameters lowered in the tissue of the hip or knee joint as well as in serum in the course of osteoarthritis?

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and more
* patient qualified for primary TKA or primary THA
* patient diagnosed with hip or knee osteoarthritis
* a complete set of tissues of good quality and volume is available
* does not meet the exclusion criteria.

Exclusion Criteria:

* lack of written consent to participate in the study or surgery
* any private or professional relationship with the Investigators
* genetic connective tissue diseases (e.g., Ehlers-Danlos syndrome and others)
* genetic metabolic diseases (e.g., gout and others)
* genetic diseases affecting the anatomy of the operated joint (e.g., dysplasia and others)
* previous surgeries altering the anatomy of the examined joint (e.g., periacetabular osteotomy, unicompartmental endoprosthesis, and others)
* patients undergoing revision after THA/TKA
* autoimmune diseases in the patient's medical history
* traumatic injury to the hip or knee joint
* previous participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary THA or TKA at the trauma and orthopedics department of the hospital in Ostrów Mazowiecka, as well as at the trauma and orthopedics department in Międzylesie Specialist Hospital in Poland.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-11-22 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Enzymatic activity of selected proteolytic enzymes in periarticular tissue homogenate (e.g., metalloproteinases and selected serine/cysteine proteases). | Perioperative/Periprocedural (during primary THA/TKA; index hospitalization)
  Enzymatic activity assessed using biochemical/spectrofluorometric methods and normalized to total protein. Each enzyme will be reported separately. Data is planned to be reported as activity units per mg protein (e.g. U/mg protein).

SECONDARY OUTCOMES:
Protein concentration of selected inflammatory markers in blood (e.g., TNF-α, IL 17α). | Perioperative/Periprocedural (day of surgery; index hospitalization for primary THA/TKA)
  Protein concentrations measured by enzyme immunoassays (EIA/ELISA). Each protein will be reported separately as pg/mL.
Trace element concentration in periarticular tissues (e.g., Zn, Cu, Fe). | Perioperative/Periprocedural (day of surgery; index hospitalization for primary THA/TKA)
  Trace element content measured by Inductively Coupled Plasma - Mass Spectrometry (ICP-MS). Each element will be reported separately. The units for serum measurements is µg/L, and for other tissue is mg/kg dry weight.
Relative mRNA expression of selected inflammatory and bone metabolism markers in periarticular tissue (e.g. TNF-α, RANK, RANKL, BMP-12, IL-17α, IL-17αR). | Perioperative/Periprocedural (day of surgery; index hospitalization for primary THA/TKA)
  Relative mRNA expression measured by RT-qPCR and reported as fold change (e.g., 2^-ΔΔCt). Each gene will be reported separately (no aggregation into a single score).

CONTACTS AND LOCATIONS:
Locations (1):
- Szpital Powiatowy im. M. Skłodowskiej-Curie, Ostrów Mazowiecka, Masovian Voivodeship, Poland